CLINICAL TRIAL: NCT06168682
Title: The Effect of Nasal Continuous Positive Airway Pressure on Oxygenation in High-risk Patients Having Gastrointestinal Endoscopy Under Deep Sedation
Brief Title: Nasal CPAP - The Treatment IMpact on Oxygenation in High-risk Patients During Deep Sedation for Endoscopy
Acronym: NAPTIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14116209135
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Continuous Positive Airway Pressure; Endoscopy; Oxygenation; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Prospective, randomized single centre trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nasal continuous positive airway pressure (Experimental): nasal continuous positive airway pressure (3-10cmH20) administered with 6 l/O2 with the SuperNO2VA™ Et produced by Vyaire Medical, Inc.
  Interventions: Device: SuperNO2VA™ Et by Vyaire Medical, Inc.
- nasal oxygen insufflation (Active Comparator): nasal oxygen insufflation with 6 l/02 will be administered as control-group/standard intervention for endoscopy
  Interventions: Device: nasal oxygen cannula

INTERVENTIONS:
Device: SuperNO2VA™ Et by Vyaire Medical, Inc. — SuperNO2VA™ Et provides a nCPAP between 3 to 10 cmH20 using a oxygenflowrate of 6l/O2
  Arms: nasal continuous positive airway pressure
Device: nasal oxygen cannula — Standard Operating Procedure (SOP) for endoscopy: Using a nasal oxygen cannula with oxygenflowrate of 6l/O2
  Arms: nasal oxygen insufflation

SUMMARY:
Deep sedation during gastrointestinal endoscopy in patients with cardiopulmonary risk factors such as respective co-morbidities or also morbid obesity is challenging. Those high-risk patients are at risk of upper airway obstruction and hypoxemia. Nasal continuous positive airway pressure may help to decrease the incidence of peri-interventional hypoxemia. However, data on nasal continuous positive airway pressure in high-risk patients having gastrointestinal endoscopy are scarce; only one randomized trial on gastroscopy in obese patients is available (Kang et al. J Anesth 2021). In a very high-risk group, namely patients assessed for heart or lung transplantation in our hospital, the risk was especially high (unpublished data).

Aim of this trial is the effect of nasal continuous positive airway pressure - compared to nasal oxygen insufflation - on the incidence of hypoxemia in high-risk patients having gastrointestinal endoscopy in deep sedation.

The investigators hypothesize that nasal continuous positive airway pressure - compared to nasal oxygen insufflation - reduces the incidence of hypoxemia in high-risk patients having gastrointestinal endoscopy in deep sedation.

DETAILED DESCRIPTION:
High risk patients were defined as American Society of Anaesthesiology (ASA) class >3 and/or BMI ≥30 kg/m², in accordance with the current World Health Organization (WHO) definition of obesity scheduled for elective gastrointestinal endoscopy with deep sedation.

The main objective was investigating the incidences of hypoxemia defined as a peripheral oxygen saturation of ≤90% registered with the monitoring system of our working station (company: Masimo; type: Root) after inducing deep sedation while under endoscopy intervention. Secondary outcomes such as the duration of the whole intervention, the duration of hypoxemia or the incidence of need for airway interventions will also be investigated.

Patients will be randomized and divided into nCPAP group and nasal oxygenation insufflation group.

Depending on the type of endoscopy a positive airway pressure between 3 and 10 cmH20 can be generated with the nCPAP mask using an oxygenflow rate of 6l/min.

Deep sedation will be performed under surveillance of an anaesthesia team using only propofol bolus adjusted to predicted body weight (PBW)(1mg/kg) followed by continuous infusion of 4mg/kg/h adjusted to lean body weight (LBW), which is described by MacDonald et al. (doi: 10.1177/1751143714565059) as :

PBW (m) (kg) = 50 + [0.91 ×(Height in cm - 152.4) PBW (f) (kg) = 45,5 + [0.91 ×(Height in cm - 152.4)

Ideal body weight (IBW) (m) (kg) = 50 + [0.9 ×(Height in cm - 154) IBW (f) (kg) = 45,5 + [0.9 ×(Height in cm - 154)

Adjusted Body Weight (ABW): IBW+0,4* (Absoluteweight-IBW)

LBW (m) (kg) = (9270 x TBW) / (6680+(216 x BMI) LBW (f) (kg) = (9270 x TBW) / (8780+(244 x BMI)

The level of sedation will be evaluated using the MOAA/S Score (modified observer's assessment of alertness/sedation scale) described by Kowalski et al. (DOI:10.1097/00003643-200706001-00097).

The sample size calculation is based on the primary outcome of the incidence of hypoxemia defined as a peripheral oxygen saturation of ≤90% after inducing deep sedation while performing endoscopy.

The incidence of the primary outcome was assumed to be 30% in nasal oxygen insufflation group and 10% in the nasal continuous positive airway pressure group. A total sample size of 158, i.e., 79 patients per group, is required to achieve 90% power in the detection of a difference of 20% between the group incidences at a significance level of 0.05 using a two-sided test of proportions. The randomization and division in subgroup "nasal continuous positive airway pressure" and "nasal oxygen insufflation" will occur prior to study entry. The entire collective will be divided into 2 populations and the allocation sealed in envelopes. The envelope will only be opened directly before the study so that investigator bias can be minimized.

ELIGIBILITY:
Inclusion Criteria:

* Adult and obese high-risk patients (ASA class ≥3 and/or BMI ≥30 kg/m², in accordance with the current WHO definition of obesity) scheduled for elective gastrointestinal endoscopy with deep sedation.

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* Cognitive impairment, that makes consent to study impossible
* Known but untreated heart disease (e.g. persistent foramen ovale (PFO), recent congestive heart failure), complicating comparability within groups

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of hypoxemia | Time between Induction of deep sedation and end of procedure (endoscopy)
  hypoxemia is defined as a peripheral oxygen saturation of ≤90% registered with the monitoring system of our working station (Phillips IntelliVue and Massimo Rad-97) after inducing deep sedation while under endoscopy intervention.

SECONDARY OUTCOMES:
Duration of intervention | Time between Induction of deep sedation and end of procedure (endoscopy)
  Total time (sec)
Duration of hypoxemia | Time between Induction of deep sedation and end of procedure (endoscopy)
  Time between hypoxemia (<90% SpO2) and recovery (> 90% SpO2) (sec)
Hypoxemic events | Time between Induction of deep sedation and end of procedure (endoscopy)
  Number of hypoxemic events per intervention/endoscopy
hypoxemia duration to procedure duration | Time between Induction of deep sedation and end of procedure (endoscopy)
  Relative ratio of hypoxemia duration compared to procedure duration
Airway intervention | Time between Induction of deep sedation and end of procedure (endoscopy)
  Incidence of airwayintervention (mask ventilation, intubation, interruption)
Sedation score | Time between Induction of deep sedation and end of procedure (endoscopy)
  Modified observer's assessment of Alertness / Sedation (MOAA/S)
Endtidal CO2 (carbon dioxide) | Time between Induction of deep sedation and end of procedure (endoscopy)
  Continuous measurement of endtidal CO2 via the mask

CONTACTS AND LOCATIONS:
Overall Officials: Karlo R Huenerbein, Dr. med., Principal Investigator — Department of Anesthesiology, Center of Anesthesiology and Intensive Care Medicine
Locations (1):
- Department of Anesthesiology, Center of Anesthesiology and Intensive Care Medicine, Hamburg, Germany

REFERENCES:
- [Derived] Hunerbein K, Sprenger C, Zollner C, de Heer J, von Wulffen M, Zimmermann K, Rosch T, Issleib M. Nasal Continuous Positive Airway Pressure to Reduce Hypoxia in Patients With Obesity Undergoing Sedated Upper Gastrointestinal Endoscopy: A Prospective Randomized Trial. Clin Gastroenterol Hepatol. 2026 Jan;24(1):113-120.e4. doi: 10.1016/j.cgh.2025.06.015. Epub 2025 Jul 1. PMID 40609816

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT06168682/Prot_SAP_000.pdf